CLINICAL TRIAL: NCT03488836
Title: Evaluation the Post Operative Pain of Endodontic Treated Molar Tooth With Race and Reciprocal Systems Among Bandarabbas Patients in 2017: A Double Blind Randomized Controlled Trial
Brief Title: Evaluation the Post Operative Pain of Endodontic Treated Molar Tooth With Race and Reciprocal Systems Among Bandarabbas Patients in 2017
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sajad Ansari Fard (Other)
Responsible Party: Sponsor-Investigator, Sajad Ansari Fard, Student, Hormozgan University of Medical Sciences
Organization: Hormozgan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 911150105
Record Dates: First submitted 2018-02-04; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- race (Active Comparator): race rotation protocol
  Interventions: Procedure: reciproc
- reciproc (Active Comparator): reciprocal endodontic treatment group
  Interventions: Procedure: race rotary

INTERVENTIONS:
Procedure: reciproc — rotary reciprocating protocol
  Arms: race
Procedure: race rotary — race rotary group protocol
  Arms: reciproc

SUMMARY:
extrusion of infected dentin into the periapical tissue has been suggested as a major source of pain after endodontic treatment. Although debris extrusion is an inevitable finding even when instrumentation is limited to the confines of the canal, different armamentarium seem to be associated with different amounts of debris extrusion. Studies on the effect of various rotary files on post-endodontic pain are very few and have yielded conflicting results with some favoring full-sequence and others leaning towards reciprocal rotary systems. This study aims at assessing the intensity of post-endodontic pain following two different rotary systems, Reciproc and race.

Methods: in this single-blind, parallel-grouped randomized clinical trial a total of 150 otherwise healthy patients aged between 20 to 50 years old with a pulpal status of irreversible pulpitis for one tooth in the upper or lower molar region were analyzed. A clinician performed the endodontic treatment in two groups, a group instrumented using race and a third group with instrumentation performed using Reciproc rotary systems.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: the otherwise healthy patients were aged between 20 to 50 years old with a pulpal status of irreversible pulpitis for one tooth in the upper or lower molar region.

Exclusion Criteria:

* Exclusion criteria: previous endodontic treatment; a history of drug intake including corticosteroids; opioids and NSAIDs in the previous 12 hours; pregnancy; complicated anatomy (curves greater than 25 degrees); calcifications; internal & external resorption; open apices; periodontal disease; swelling & abscess; presence of periapical lesions; sensitivity to percussion and lack of occlusal contact.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-05-02 (Estimated); Primary Completion 2018-07-02 (Estimated); Study Completion 2018-11-02 (Estimated)

PRIMARY OUTCOMES:
change of the Visual analogue scale | 6-12-18-24-48-72 hours
  change of the vas evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Dental clinic of BandarAbbas faculty of dentistry, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: Undecided